CLINICAL TRIAL: NCT07239128
Title: Efficacy of Low-Level Light Therapy in Combination With Topical Non-Steroidal Immunosuppressants for the Treatment of Dry Eye Disease
Brief Title: Photobiomodulation in Combination With Topical Cyclosporine A or Tacrolimus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Centro Oculistico Borroni (Other)
Responsible Party: Principal Investigator, Antonio Ballesteros Sánchez, OD, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 29/20092016
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Dry Eye Disease (DED)
Keywords: Topical Cyclosporine A; Topical Tacrolimus; Low-level light therapy
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Low-Level Light Therapy; Cyclosporine; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Active-controlled (CsA and Tacrolimus)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were masked to CsA and Tacrolimus, but not to LLLT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CsA (Active Comparator): CsA 0.1% twice per day
  Interventions: Drug: Topical Cyclosporine A
- Tacrolimus (Active Comparator): Tacrolimus 0.1% twice per day
  Interventions: Drug: Topical tacrolimus
- LLLT-CsA (Experimental): Three 15-minute sessions of LLLT were performed at weekly intervals. The treatment was delivered with a wavelength of 625 nm and a radiance of 35 mW/cm², resulting in a total energy dose of approximately 32 J/cm² applied to the facial and eyelid regions with eyes closed.
  CsA 0.1% twice per day.
  Interventions: Device: Low-level light therapy (LLLT); Drug: Topical Cyclosporine A
- LLLT-Tacrolimus (Experimental): Three 15-minute sessions of LLLT were performed at weekly intervals. The treatment was delivered with a wavelength of 625 nm and a radiance of 35 mW/cm², resulting in a total energy dose of approximately 32 J/cm² applied to the facial and eyelid regions with eyes closed.
  Tacrolimus 0.1% twice per day.
  Interventions: Device: Low-level light therapy (LLLT); Drug: Topical tacrolimus

INTERVENTIONS:
Device: Low-level light therapy (LLLT) — Three 15-minute sessions were performed at weekly intervals. The treatment was delivered with a wavelength of 625 nm and a radiance of 35 mW/cm², resulting in a total energy dose of approximately 32 J/cm² applied to the facial and eyelid regions with eyes closed.
  Other Names: Photobiomodulation
  Arms: LLLT-CsA; LLLT-Tacrolimus
Drug: Topical Cyclosporine A — CsA 0.1% twice per day
  Arms: CsA; LLLT-CsA
Drug: Topical tacrolimus — Tacrolimus 0.1% twice per day
  Arms: LLLT-Tacrolimus; Tacrolimus

SUMMARY:
The objective of the study is to evaluate the effectiveness of Low-level light therapy (LLLT) in combination with either topical Cyclosporine A (CsA) or topical Tacrolimus, using each non-steroidal immunosuppressant as an active control.

ELIGIBILITY:
Inclusion Criteria:

(1) Ocular Surface Disease Index (OSDI) score > 13; (2) non-invasive tear film break-up time (NIBUT) < 10 seconds; and (3) tear meniscus height < 0.25 mm.

Exclusion Criteria:

(1) structural abnormalities of the eyelids; (2) active blepharitis; (3) corneal disorders that could interfere with study assessments, such as active corneal infections or corneal dystrophies; (4) active ocular allergy; (5) history of procedures for DED treatment within the previous 12 months, such as eyelid exfoliation, thermal eyelid therapies, light therapies, or quantum molecular resonance (QMR); (6) history of intraocular or laser ocular surgery within the past 5 years; (7) current use of topical antibiotics or anti-inflammatory agents; (8) diagnosis of systemic autoimmune disease; (9) contact lens wear; (10) pregnancy or lactation; and (11) inability to understand or provide informed consent.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index (OSDI) | From baseline visit to the end of follow-up (12 months)
  A standardized questionnaire designed to assess the symptoms of dry eye disease and their impact on vision-related functioning. It consists of 12 items that evaluate the frequency of symptoms, environmental triggers, and functional limitations over the previous week. The OSDI provides a score from 0 to 100, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Non-invasive tear film break-up time (NIBUT) | From baseline visit to the end of follow-up (12 months)
  NIBUT is a clinical test used to evaluate tear film stability without the use of dyes. It measures the time interval between a complete blink and the first appearance of a disruption or break in the tear film. Shorter NIBUT values indicate reduced tear film stability.
Tear meniscus height (TMH) | From baseline visit to the end of follow-up (12 months)
  TMH is a quantitative parameter used to assess tear volume. Reduced TMH values are indicative of aqueous tear deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Borroni, MD, PhD, Principal Investigator — Department of Ophthalmology, Riga Stradins University, Riga, Latvia; Antonio Spinelli, MD, Principal Investigator — Biomeeting Day Surgery center
Locations (2):
- Italy (2):
  - Biomeeting Day Surgery center, Reggio Calabria, Calabria
  - Centro Oculistico Borroni, Gallarate, Varese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones L, Craig JP, Markoulli M, Karpecki P, Akpek EK, Basu S, Bitton E, Chen W, Dhaliwal DK, Dogru M, Gomes JAP, Koehler M, Mehta JS, Perez VL, Stapleton F, Sullivan DA, Tauber J, Tong L, Trave-Huarte S, Wolffsohn JS; TFOS Collaborator Group. TFOS DEWS III: Management and Therapy. Am J Ophthalmol. 2025 Nov;279:289-386. doi: 10.1016/j.ajo.2025.05.039. Epub 2025 Jun 2. PMID 40467022
- [Background] Antwi A, Schill AW, Redfern R, Ritchey ER. Effect of low-level light therapy in individuals with dry eye disease. Ophthalmic Physiol Opt. 2024 Nov;44(7):1464-1471. doi: 10.1111/opo.13371. Epub 2024 Aug 2. PMID 39096028
- [Background] Moawad P, Shamma R, Hassanein D, Ragab G, El Zawahry O. Evaluation of the effect of topical tacrolimus 0.03% versus cyclosporine 0.05% in the treatment of dry eye secondary to Sjogren syndrome. Eur J Ophthalmol. 2022 Jan;32(1):673-679. doi: 10.1177/1120672121992680. Epub 2021 Feb 2. PMID 33530719

DOCUMENTS (2):
  • Study Protocol (2025-10-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT07239128/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT07239128/SAP_001.pdf